CLINICAL TRIAL: NCT00737152
Title: Phase II, Open-Label Study to Assess the Cardiovascular Side Effects and Efficacy for Reducing Blood Glucose Level in Type II Diabetes Mellitus Patients Being Treated With RAS 130 With or Without Diet and Exercise
Brief Title: Evaluate the Side Effects and Benefits of RAS 130 With or Without Diet and Exercise in Type II Diabetes Mellitus
Acronym: ASI-DMII
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: American Scitech International (Other)
Collaborators: Proactive Clinical Research (Unknown)
Responsible Party: Dr. Ratna Grewal, American Scitech International
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASI-DMII 0808
Record Dates: First submitted 2008-08-14; First posted 2008-08-18 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Type II Diabetes Mellitus
Keywords: RAS 130; Exercise; Diabetes Mellitus; Type II Diabetes; Diabetes; Aerobic
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity; Diabetes Mellitus | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): All subjects will take RAS 130 administered orally in tablet form at a starting dose of 4 mg once a day or 2 mg tablets twice a day.
  Interventions: Other: RAS 130 with diet and exercise

INTERVENTIONS:
Other: RAS 130 with diet and exercise — Entire population, which will also include existing patients, will be treated with RAS 130 along with diet and exercise. By the end of 6 months: 3 months of study and 3 months of follow-up, the entire population will be divided into two groups which will be determined through endpoints. The first group will be subjects with diet and exercise and the second group will be subjects without diet and exercise. The endpoints for the division of the groups are given in the design of the study.
  Other Names: diet and exercise

SUMMARY:
Rationale: RAS 130 is an anti-diabetic agent used to lower the blood glucose level in Type II Diabetes mellitus (non-insulin-dependent diabetes) patients with proper diet and exercise. RAS 130 works by restoring proper response to insulin in the body. RAS 130 acts primarily by increasing insulin sensitivity which improves glycemic index. It is presumed that RAS 130 does not cause cardiovascular side effects if it is given to Type II diabetes mellitus patients leading a healthy life style. Specifically, controlling diet is done according to American Diabetic Association & American Heart Association guidelines and also through doing aerobic exercises. Guideline for aerobic exercise is given in the design of the study.

Exercise is helpful in controlling body weight which can lower the risk for heart disease. Diabetes itself is one of the compounding factors for heart diseases. Exercise helps lowering the LDL cholesterol and raising the HDL cholesterol which is required to prevent heart diseases and achieve a better quality of life.

Purpose: The aim of this study is to prospectively assess and evaluate the cardiovascular side effects and reduction of blood glucose levels in the Type II Diabetes mellitus patients treated with RAS 130, who either met, or failed to meet criteria for diet and exercise.

DETAILED DESCRIPTION:
Objectives:

Primary Objective:

To determine the relatedness of cardio toxicity as a side effect in subjects with DM II who are treated with RAS 130 who either met, or failed to meet the criteria for diet and exercise.

Hypothesis I: There will be no evidence of cardiovascular side effects in subjects who are determined to have maintained proper diet and exercise "healthy lifestyle" throughout the study.

Hypothesis II: There may be evidence of cardiovascular side effects in subjects who are determined to neglect proper diet and exercise "unhealthy lifestyle" throughout the study.

Secondary Objective:

To determine the effectiveness of RAS 130 on the reduction of blood glucose levels in subjects with DM II.

Hypothesis III: RAS 130 will be effective in reducing blood glucose levels as a single agent.

Hypothesis IV: RAS 130 will be effective in reducing blood glucose in combination with other anti- diabetic agents.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Type II Diabetes Mellitus (non-insulin-dependent), not taking any anti-diabetic agent.
2. Fasting blood glucose level below 250mg/dL
3. Age 30 to 60 years
4. Both genders
5. HbA1c of 6.0% to 13.0%, inclusive
6. Body mass index (BMI) below 40 kg/m2
7. Female subjects not pregnant, not lactating, post-menopausal, surgically sterile or using effective contraceptive measures are included.
8. Provide signed Informed Consent

Exclusion Criteria:

1. Subject unable to give Informed Consent
2. Patients with Type I Diabetes Mellitus

   a. History of ketoacidosis
3. Serum creatinine > 2.0 mg or above
4. Liver Function Test; Elevated liver enzymes: ALT/AST (2.5 times the upper limit of the reference range), Bilirubin Testing - Accept three fold, A/G ratio - Accept two fold
5. Hypercholesterolemia (more than 300mg)
6. Myocardial Infarction (MI) within 6 months
7. Severe or unstable angina
8. Elevated triglycerides >500 mg/dL
9. Abnormal EKG reading
10. Abnormal assessment in stress Echocardiography (ultrasound imaging)for Left Ventricular ejection fraction for congestive heart failure
11. Anemia (Hb <11 g/dl for men or <10 g/dl for women)
12. Blood Dyscrasia, Decrease in Hematocrit - Accept two fold, Low WBC count - Accept one fold, Decrease platelet count - Accept three fold
13. Macular edema/ macular degeneration
14. Patients who are taking insulin
15. Subjects with systolic blood pressure >170 mmHg or diastolic blood pressure >90 mmHg
16. Active participation in another trial
17. Subject physically unable to perform exercise due to neurologic or orthopedic conditions.
18. Patients taking antipsychotic medications.
19. Subjects testing positive for the illicit drugs (cocaine, amphetamines, heroin)
20. Subjects who smoke tobacco products
21. Females who are lactating, pregnant, or planning to become pregnant
22. Signs and symptoms of Congestive heart failure (such as shortness of breath or swelling in upper extremities)
23. History of severe edema or a medically serious fluid retention

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 460 (Estimated)
Dates: Start 2011-07; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
To determine cardiovascular side effects such as coronary artery disease (CAD) and congestive heart failure (CHF) in patients treated with RAS 130 along with diet and exercise. | 6 months

SECONDARY OUTCOMES:
To determine the effect of RAS 130 on reduction of blood glucose level with or without diet and exercise | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ratna Grewal, MD, Study Chair — American Scitech International - eCRO; Prem Nandiwada, MD, Principal Investigator — Raritan Bay Medical Center
Locations (5):
- United States (3):
  - MedCenter, East Brunswick, New Jersey
  - Robertwood Johnson Hospital, New Brunswick, New Jersey
  - Raritan Bay Medical Center, Perth Amboy, New Jersey
- India (2):
  - Sri Ramachandra University, Porur, Chennai
  - Dr. JL Rohatagi Hospital, Sarvoday Nagar, Kanpur, Uttar Pradesh